CLINICAL TRIAL: NCT05657210
Title: Does KRAS Codon 13 Mutation Have Prognostic Value in Colorectal Cancer?
Brief Title: Prognostic Value of Each Codon-specific KRAS Mutation in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Duck-Woo Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2203-742-101
Record Dates: First submitted 2022-12-10; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Mutation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- KRAS wildtype
- KRAS codon 12 mutation
  Interventions: Genetic: Mutation
- KRAS codon 13 mutation
  Interventions: Genetic: Mutation
- KRAS codon 61 mutation
  Interventions: Genetic: Mutation

INTERVENTIONS:
Genetic: Mutation
  Groups: KRAS codon 12 mutation; KRAS codon 13 mutation; KRAS codon 61 mutation

SUMMARY:
This retrospective study reviewed 3,144 patients who underwent surgery for colorectal cancer. This study was designed to comprehend the clinicopathological characteristics associated with individual codon-specific KRAS mutations in colorectal cancer.

DETAILED DESCRIPTION:
This study was designed to comprehend the clinicopathological characteristics associated with individual codon-specific KRAS mutations in colorectal cancer including codon 12, 13, and 61. Furthermore, the main objective of this study was to determine whether KRAS codon 13 mutation could serve as a prognostic biomarker of colorectal cancer in a relatively large cohort of subjects. Overall survival (OS) and recurrence-free survival (RFS) were calculated from the date of surgery and compared using the Kaplan-Meier method and log-rank test. For analysis of risk factors for tumor recurrence, Cox proportional hazards regression model was used with the covariance input criterion set as < 0.1. Patients were subdivided based on primary tumor location (colon versus rectum), and MSI status (MSS/MSI-low versus MSI-high).

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent surgery for colorectal cancer from January 2009 to December 2019.

Exclusion Criteria:

* incomplete data on KRAS mutation
* incomplete data on microsatellite instability (MSI) status
* dual or triple KRAS mutation
* stage IV

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Three tertiary referral hospitals between January 2009 to December 2019
Sampling Method: Probability Sample
Enrollment: 2203 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
5-year Recurrence-free survival (RFS) of KRAS wildtype and each codon-specific KRAS mutation | from the date of surgery to the event(recurrence and death) up to 5 years
5-year Overall survival (OS) of KRAS wildtype and each codon-specific KRAS mutation | from the date of surgery to the event(death) up to 5 years

SECONDARY OUTCOMES:
Recurrence-related factor | Recurrence in 5 years after the date of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No